CLINICAL TRIAL: NCT04910685
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2/3 Study of BLU-263 in Indolent Systemic Mastocytosis
Brief Title: (HARBOR) Study to Evaluate Efficacy and Safety of BLU-263 Versus Placebo in Patients With Indolent Systemic Mastocytosis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLU-263-1201
Record Dates: First submitted 2021-05-17; First posted 2021-06-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Indolent Systemic Mastocytosis; Smoldering Systemic Mastocytosis
Keywords: ISM; SSM
MeSH Terms: conditions — Mastocytosis, Systemic

STUDY DESIGN:
Intervention Model Description: Part 1 and Part 2: Randomized, Blinded Part 3, Part K, Part S and PK groups: Non-randomized, Open-label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- (Part 1) Elenestinib Dose 1 + SDT (Experimental): Participants will receive SDT and elenestinib. SDT will be determined on a per participant basis. Elenestinib will be administered orally, once daily until completion of Part 1.
  Interventions: Drug: Elenestinib
- (Part 1) Elenestinib Dose 2 + SDT (Experimental): Participants will receive SDT and elenestinib. SDT will be determined on a per participant basis. Elenestinib will be administered orally, once daily until completion of Part 1.
  Interventions: Drug: Elenestinib
- (Part 1) Elenestinib Dose 3 + SDT (Experimental): Participants will receive SDT and elenestinib. SDT will be determined on a per participant basis. Elenestinib will be administered orally, once daily until completion of Part 1.
  Interventions: Drug: Elenestinib
- (Part 1) Placebo + SDT (Placebo Comparator): Participants will receive SDT and matching placebo. SDT will be determined on a per participant basis. Placebo will be administered orally, once daily until completion of Part 1.
  Interventions: Drug: Placebo
- (Part 2) Elenestinib Dose 1 + SDT (Experimental): Participants will receive SDT and elenestinib. SDT will be determined on a per participant basis. Elenestinib will be administered orally, once daily for approximately 48 weeks.
  Interventions: Drug: Elenestinib
- (Part 2) Placebo + SDT (Placebo Comparator): Participants will receive SDT and matching placebo. SDT will be determined on a per participant basis. Placebo will be administered orally, once daily for approximately 48 weeks.
  Interventions: Drug: Placebo
- (Part 3) Elenestinib + SDT (Experimental): Participants will receive SDT and elenestinib. SDT will be determined on a per participant basis. Elenestinib will be administered orally, once daily for up to approximately 5 years.
  Interventions: Drug: Elenestinib
- (Part S) Elenestinib Dose 1 + SDT (Experimental): Participants will receive SDT and elenestinib. SDT will be determined on a per participant basis. Elenestinib will be administered orally, once daily for up to approximately 5 years.
  Interventions: Drug: Elenestinib
- (Part K) Elenestinib Dose 1 + SDT (Experimental): Participants will receive SDT and elenestinib. SDT will be determined on a per participant basis. Elenestinib will be administered orally, once daily for up to approximately 5 years.
  Interventions: Drug: Elenestinib
- (PK groups) Elenestinib + SDT (Experimental): Participants will receive SDT and elenestinib. SDT will be determined on a per participant basis. Elenestinib will be administered orally, once daily for up to approximately 5 years.
  Interventions: Drug: Elenestinib

INTERVENTIONS:
Drug: Elenestinib — Elenestinib oral tablet
  Other Names: BLU-263
  Arms: (PK groups) Elenestinib + SDT; (Part 1) Elenestinib Dose 1 + SDT; (Part 1) Elenestinib Dose 2 + SDT; (Part 1) Elenestinib Dose 3 + SDT; (Part 2) Elenestinib Dose 1 + SDT; (Part 3) Elenestinib + SDT; (Part K) Elenestinib Dose 1 + SDT; (Part S) Elenestinib Dose 1 + SDT
Drug: Placebo — Placebo oral tablet
  Arms: (Part 1) Placebo + SDT; (Part 2) Placebo + SDT

SUMMARY:
This is a randomized, double-blind, placebo-controlled, Phase 2/3 study comparing the efficacy and safety of elenestinib (BLU-263) + symptom directed therapy (SDT) with placebo + SDT in participants with indolent systemic mastocytosis (ISM) whose symptoms are not adequately controlled by SDT. Parts 1 and 2 will enroll participants with ISM. Participants enrolled in Part 2 will roll over onto Part 3 to receive treatment with elenestinib in an open-label fashion following completion of the earlier Part. Part K will enroll participants with ISM who have previously received an approved selective KIT inhibitor. The study also includes pharmacokinetic (PK) groups that will enroll participants with ISM.

ELIGIBILITY:
Key Inclusion Criteria:

All Participants:

-Participant must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2.

Part 1 and PK groups:

* Participant has confirmed diagnosis of ISM, confirmed by Central Pathology Review
* Participant must have failed to achieve adequate symptom control for 1 or more Baseline symptoms, as determined by the Investigator, with at least 2 of the following symptom-directed therapies administered: H1 blockers, H2 blockers, proton-pump inhibitors, leukotriene inhibitors, cromolyn sodium, corticosteroids, or omalizumab.
* Participants must have SDT for ISM symptom management stabilized for at least 14 days prior to starting screening procedures.
* For participants receiving corticosteroids, the dose must be ≤ 20 mg/day prednisone or equivalent, and the dose must be stable for ≥ 14 days.

Part K:

-Participant has confirmed diagnosis of ISM, confirmed by Central Pathology Review

Part S:

-Participant has confirmed diagnosis of SSM, confirmed by Central Pathology Review of BM biopsy and central review of B- and C-findings by WHO diagnostic criteria.

Part 2:

-Participant has confirmed diagnosis of ISM, confirmed by Central Pathology Review

Key Exclusion Criteria:

* Participant has been diagnosed with any of the following WHO systemic mastocytosis (SM) sub-classifications: cutaneous mastocytosis only, SM with an associated hematologic neoplasm of non-MC lineage (SM-AHN), aggressive SM, mast cell leukemia, or mast cell sarcoma.
* Participant has been diagnosed with another myeloproliferative disorder.
* Participant has organ damage attributable to SM.
* Participant has clinically significant, uncontrolled, cardiovascular disease
* Participant has a QT interval corrected using Fridericia's formula (QTcF) > > 470 milliseconds (msec) (for females) or > 450 msec (for males).
* Participant has a history of a primary malignancy that has been diagnosed or required therapy within 3 years. The following prior malignancies are not exclusionary: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate cancer, and completely resected carcinoma in situ of any site.
* Time since any cytoreductive therapy including masitinib and midostaurin should be at least 5 half-lives or 14 days (whichever is longer), and for cladribine, interferon alpha, pegylated interferon, or antibody therapy < 28 days or 5 half-lives of the drug (whichever is longer), before beginning the screening period.
* Participant has received radiotherapy or psoralen and ultraviolet A (PUVA) therapy < 14 days before beginning the screening period.

Other protocol-defined criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2032-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 12 weeks
Part 1: Mean change from baseline in ISM-Symptom in Assessment Form (ISM-SAF) Total Symptom Score (TSS) | Baseline, Week 13
Part 2: Mean change from baseline in ISM-SAF TSS | Baseline, Week 49
Part 3: Number of participants with Adverse Events (AEs) | Up to 5 years
Part 3: Change from baseline in ISM-SAF TSS | Baseline up to 5 years

SECONDARY OUTCOMES:
Part 1: Change from baseline in serum tryptase | Baseline, Week 13
Part 1: Change from baseline in KIT D816V allele fraction in blood | Baseline, Week 13
Part 1: Change from baseline in Bone Marrow (BM) mast cells | Baseline, Week 13
Part 1: Mean change from baseline in ISM-SAF individual symptom scores | Baseline, Week 13
Part 1: Time to achieve 30% reduction from baseline in ISM-SAF TSS | Baseline up to Week 13
Part 1: Time to achieve 30% reduction from baseline in ISM-SAF domain scores | Baseline up to Week 13
Part 2: Proportion of participants achieving normalized tryptase | Baseline up to Week 49
Part 2: Proportion of participants who achieve an undetectable level or at least a 50% reduction in KIT D816V Variant Allele Frequency (VAF) | Baseline up to Week 49
Part 2: Proportion of participants achieving symptom control as defined by achieving mild symptoms | Baseline up to Week 49
Part 2: Mean percent change from baseline in Bone Mineral Density (BMD) | Baseline, Week 49
Part 2: Mean change from baseline in the annualized rate of anaphylaxis events | Baseline, Weeks 25 to 48
Part 2: Mean change from baseline in Quality of Life (QoL) scores | Baseline, Week 49
Part 2: Mean change from baseline in ISM-SAF domain scores | Baseline, Week 49
Part 2: Number of participants with AEs | Up to Week 49
Part 2: Proportion of participants with a 50% reduction in ISM-SAF TSS | Baseline, Weeks 24 and 48
Part 2: Proportion of participants with a 50% reduction in ISM-SAF domain scores | Baseline, Weeks 24 and 48
Part 2: Proportion of participants with a 30% reduction in ISM-SAF TSS | Baseline, Weeks 24 and 48
Part 2: Proportion of participants with a 30% reduction in ISM-SAF domain scores | Baseline, Weeks 24 and 48
Part 3: Proportion of participants achieving symptom control as defined by achieving mild symptoms | Baseline up to 5 years
Part 3: Change from baseline in ISM-SAF domain scores | Baseline, up to 5 years
Part 3: Proportion of participants achieving a normalized tryptase | Baseline up to 5 years
Part 3: Change from baseline in BMD | Baseline up to 5 years
Part 3: Change from baseline in the annualized rate of anaphylaxis events | Baseline up to 5 years
Parts 2 and 3: Change from baseline in serum tryptase | Baseline up to 5 years
Parts 2 and 3: Change from baseline in KIT D816V allele fraction in blood | Baseline up to 5 years
Parts 2 and 3: Change from baseline in Bone Marrow (BM) mast cells | Baseline up to 5 years
Parts 2 and 3: Proportion of participants achieving controlled disease | Baseline up to 5 years
Parts 2 and 3: Change from baseline in skin lesions as assessed by the fractional body surface area of the most affected skin area | Baseline up to 5 years
Parts 2 and 3: Change from baseline in the number of concomitant medications identified as SDT | Baseline up to 5 years
Parts 2 and 3: Change from baseline in ISM-SAF Individual Symptom Scores | Baseline up to 5 years
Parts 2 and 3: Change from baseline in ISM-SAF Lead (most severe) Symptom Score | Baseline up to 5 years
Parts 2 and 3: Change from baseline in QoL scores | Baseline up to 5 years
Part S: Number of participants with AEs | Baseline up to 5 years
Part S: Proportion of participants who achieve a Pure Pathologic Response (PPR) | Baseline up to 5 years
Part S: Mean change from baseline in ISM-SAF | Baseline, Week 25
Part K: Number of participants with AEs | Baseline up to 5 years
Part K: Change from baseline in serum tryptase | Baseline up to 5 years
Part K: Change from baseline in KIT D816V allele fraction in blood | Baseline up to 5 years
Part K: Mean change from baseline in ISM-SAF TSS | Baseline up to 5 years
Part K: Change from baseline in QoL scores | Baseline up to 5 years

CONTACTS AND LOCATIONS:
Locations (54):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford Cancer Institute, Palo Alto, California
  - UCHealth Blood Disorders and Cell Therapies Center - Anschutz Medical Campus, Aurora, Colorado
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Medicine University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
- Australia (2):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- Kepler Universitatsklinikum, Med Campus III. Clinic of Internal Medicine 3 - Hematology and Oncology, Linz, Austria
- Unitversitair Ziekenhuis Antwerpen, Edegem, Antwerpen, Belgium
- France (9):
  - CHU Amiens-Picardie, Amiens
  - CHU de Caen, Caen
  - CHU Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - CHU de Nantes, Nantes
  - Hôpital de la Pitié Salpétrière, Paris
  - Hôpital Necker - Départementd 'HématologieA dultes, Paris
  - CHU de Poitiers, Poitiers
  - CHU Toulouse - Hopital Larrey, Toulouse
- Germany (6):
  - Universitätsklinikum RWTH Aachen Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzelltransplantation, Aachen
  - Charité - Universitätsmedizin Berlin Institute of Allergology, Berlin
  - University Clinic Erlangen, Erlangen
  - University Clinic Hamburg Eppendorf, Hamburg
  - Universitätsmedizin Mannheim III. Medizinische Klinik Universität Heidelberg Medizinische Fakultät Mannheim, Mannheim
  - LMU Klinikum, Munich
- Italy (7):
  - UOC Ematologia, Milan, Lombardy
  - SOD Ematologia (Ambulatori)- AOUC Azienda Ospedaliero Universitaria Careggi, Florence, Tuscany
  - Unita Operativa di Ematologia AOU Policlinico S. Orsola-Malpighi, Bologna
  - AOU Policlinico G.Rodolico - San Marco, Catania
  - S.C. Ematologia Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - S.S.D. Immunologia Clinica e Allergologia Azienda Ospedaliera Universitaria San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Unità Operativa di Allergologia Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Netherlands (2):
  - ErasmusMC, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen
- Oslo University Hospital, Oslo, Norway
- Portugal (3):
  - Centro Hospitalar de Lisboa Central, E.P.E. - Hospital de Santo Antonio dos Capuchos, Lisbon
  - CHUPorto, EPE - Hospital de Santo António, Porto
  - Centro Hospitalar Universitario Sao Joao, E.P.E., Porto
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Virgen del Valle - Instituto de Estudios de Mastocitosis de Castilla-La Mancha, Toledo
- Uppsala University Hospital, Uppsala, Sweden
- Switzerland (2):
  - University Hospital Basel, Basel
  - Luzerner Kantonsspital, Lucerne
- United Kingdom (5):
  - University Hospital of Wales, Cardiff, Wales
  - University Hospital of Wales, Cardiff
  - Guy's and St Thomas's NHS Foundation Trust, London
  - Cancer and Haematology Centre, Oxford
  - University Hospital Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No